CLINICAL TRIAL: NCT04136223
Title: BERTHA Study: Rheumatoid Arthritis-Associated Interstitial Lung Disease: Characterization of Lung Disease Progression. A Multicenter, Observational Study
Brief Title: Rheumatoid Arthritis-Associated Interstitial Lung Disease: Characterization of Lung Disease Progression
Acronym: BERTHA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital do Coracao (Other)
Collaborators: Bristol-Myers Squibb (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: BERTHA_IM101-839
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Lung; Rheumatoid Arthritis; Interstitial Lung Disease; Pulmonary Fibrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA-ILD: Consecutive adult patients (aged >18 years) with RA* and interstitial lung disease
  *in accordance with the American College of Rheumatology (ACR) classification criteria of 2010

SUMMARY:
BERTHA study´s primary objective is to characterize Rheumatoid Arthritis-associated Interstitial Lung Disease (RA-ILD) progression and to define a combination of biomarkers, genetic and clinical variables capable of identifying patients at risk of RA-ILD progression

DETAILED DESCRIPTION:
BERTHA is a multicentric, observational study that will enroll 100 RA-ILD patients to be followed for 2 years.

Interstitial Lung Disease (ILD) progression will be ascertained by quantitative image analysis and functional parameters. Variables associated with progression with be identified.

Additionally, RA-ILD endotypes will be investigated as well as their association with RA-ILD progression.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive adult patients (aged >18 years) meeting RA diagnostic criteria in accordance with ACR 2010
2. Presence of interstitial lung disease 2.1 ILD Definition: presence of interstitial alterations in HRCT associated to functional derangements and/or symptoms
3. Patient agrees with having follow-up visits every 6 months for 2 years

Exclusion Criteria:

1. Pregnancy or intending to become pregnant
2. Overlap with other diseases that occurs with ILD (other collagenoses, vasculitis, inflammatory bowel disease)
3. Presence of advanced ILD, characterized by:

   a. Dyspnea rated as modified Medical Research Council 4 (mMRC4) on routine visit
4. Presence of significant Arterial Pulmonary Hypertension:

   1. Evidence of Right ventricular failure evidence by echocardiography
   2. Previous right chamber catheterism showing cardiac index < 2 liters/min/m²
5. Significant co-morbidity impacting respiratory system (e.g., congestive heart failure, lung neoplasm, active tuberculosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA-ILD patients defined by altered imaging and associated functional derangements and/ or symptoms
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Interstitial Lung Disease progression - FVC | 2 years
  FVC longitudinal behavior (continuous variable)

SECONDARY OUTCOMES:
Interstitial Lung Disease progression - imaging | 2 years
  quantitative overall disease progression (continuous variable) & %VRS (vessel related structures) > 4.4% if access to CALIPER software
Interstitial Lung Disease progression - death | 2 years
  Time to death or lung transplant
Interstitial Lung Disease progression - FVC dichotomous variable | 2 years
  Proportion of patients with a change from baseline in the %Forced Vital Capacity (FVC):
  1. greater or equal to 10% or
  2. between 5 and 10% and worsening of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Alexandra Latini, PhD, Study Chair — Federal University of Santa Catarina; Leticia Kawano-Dourado, MD, Study Chair — HCOR Research Institute, Hospital do Coracao, São Paulo, Brazil
Locations (5):
- Brazil (5):
  - Hospital Universitário de Brasilia (HUB), Brasília, Federal District
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
  - Universidade Estadual de Campinas (UNICAMP), Campinas
  - LABOX - Federal University of Santa Catarina (UFSC), Florianópolis
  - LAPOGE - Federal University of Santa Catarina (UFSC), Florianópolis

IPD SHARING:
Plan to Share IPD: Yes
Under development
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code